CLINICAL TRIAL: NCT04835649
Title: The Effectiveness of Task-Oriented Training Based Telerehabilitation in Improving Upper Extremity Motor Function in Parkinson's Patients
Brief Title: The Effectiveness of Telerehabilitation in Improving Upper Extremity in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1- PD- UE-Telerehabilitation
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Telerehabilitation; Task-oriented; upper extremity
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups as exercise group and control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The group that will receive task-oriented training via telerehabilitation
  Interventions: Other: Exercise
- Control group (Placebo Comparator): The control group only will be given a home program that includes walking and balance exercises
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both groups will receive exercise-based training

SUMMARY:
Parkinson's Disease (PD) is a disease that affects the functional skills of the upper extremity with clinical findings such as bradykinesia, rigidity, and hypokinesia and causes limitations in the daily life activities of the patients. Task-oriented training (TOT) is a highly individualized, client-centered, occupational therapy, functional-based intervention compatible with motor learning and motor control principles such as intensive motor training, variable practice, and intermittent feedback. Few studies have been found on the TOT of the upper extremity in PD. Telerehabilitation of Parkinson's patients shows many strengths, such as cost-related and time-dependent ease, and the possibility of telecommunication with clinicians. In addition, the refinement of digital health solutions with the goal to offer a patient-tailored intervention remains an ongoing process. There are a limited number of studies on TOT and telerehabilitation of the upper extremity in PD. In addition, no studies have been found applying TOT through telerehabilitation. For this purpose, a study including TOT-based telerehabilitation in upper extremity education in PD was planned.

DETAILED DESCRIPTION:
This study is a randomized controlled study. The patients will be randomly divided into two groups as exercise and control. Balance and walking exercises consisting of 3 days a week for 6 weeks will be given to both groups as a home program. In addition, the exercise group will receive TOT-based telerehabilitation via video conferencing 3 days a week for 6 weeks. TOT will be formed from daily life activities such as reaching out, grasping, writing, and manual skills, which are frequently used in daily life. As the outcome measures, disease severity and disability, finger and hand function, hand strength, and quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 45- 70 years of age
* Having diagnosed with "Parkinson's Disease" by a specialist physician
* Having between 1-3 stages according to the Hoehn and Yahr Scale
* Mini-Mental Test score more than or equal 24

Exclusion Criteria:

- Any orthopedic, vision, hearing, cardiovascular, or perception problems that may affect the research results

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Manual dexterity performance - Baseline | Assessment will be conducted before the intervention
  Nine Hole Peg test (9-HPT)
Manual dexterity performance - Post intervention | Assessment will be conducted immediately after the intervention
  Nine Hole Peg test (9-HPT)
Finger and hand function - Baseline | Assessment will be conducted before the intervention
  Jebsen-Taylor Hand Function Test (JTHFT)
Finger and hand function - Post intervention | Assessment will be conducted immediately after the intervention
  Jebsen-Taylor Hand Function Test (JTHFT)
Upper extremity performance (coordination, dexterity and functioning) - Baseline | Assessment will be conducted before the intervention
  Action Research Arm Test (ARAT)
Upper extremity performance (coordination, dexterity and functioning) - Post intervention | Assessment will be conducted immediately after the intervention
  Action Research Arm Test (ARAT)

SECONDARY OUTCOMES:
Isometric hand strength - Baseline | Assessment will be conducted before the intervention
  J-Tech ™
Isometric hand strength - Post intervention | Assessment will be conducted immediately after the intervention
  J-Tech ™
Isometric pinch strength - Baseline | Assessment will be conducted before the intervention
  Baseline® pinch meter
Isometric pinch strength - Post intervention | Assessment will be conducted immediately after the intervention
  Baseline® pinch meter
Disease severity and disability - Baseline | Assessment will be conducted before the intervention
  MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The MDS-UPDRS has a maximum score of 272 and is composed of four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications) (UPDRS). (0= best , 272= worst)
Disease severity and disability - Post intervention | Assessment will be conducted immediately after the intervention
  MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The MDS-UPDRS has a maximum score of 272 and is composed of four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications) (UPDRS). (0= best , 272= worst)
Health-related Quality of Life - Baseline | Assessment will be conducted before the intervention
  Parkinson's Disease Questionnaire 8 (PDQ-8). There are 8 questions in total and each question is scored from 0-4 points. High score indicates decreased quality of life
Health-related Quality of Life - Post intervention | Assessment will be conducted immediately after the intervention
  Parkinson's Disease Questionnaire 8 (PDQ-8). There are 8 questions in total and each question is scored from 0-4 points. High score indicates decreased quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sefa Eldemir, PT, MSc., Study Chair — Research Assistant; Arzu Güçlü-Gündüz, PT, PhD., Study Director — Professor
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- See also: Related info — https://pubmed.ncbi.nlm.nih.gov/28578819/
- See also: Related info — https://pubmed.ncbi.nlm.nih.gov/32117009/